CLINICAL TRIAL: NCT05097885
Title: Pilot Investigation on the Health Benefits of Sub Acute (12 Week) Whole-body Vibration Training
Brief Title: Health Benefits of Whole-body Vibration
Acronym: VIBE-Rx
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Ryan Harris, Professor, Augusta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1818010
Record Dates: First submitted 2021-10-15; First posted 2021-10-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Whole-body Vibration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sub Acute (12 week) Whole Body Training (Experimental)
  Interventions: Other: Sub Acute Whole Body Vibration Training

INTERVENTIONS:
Other: Sub Acute Whole Body Vibration Training — Participants will be given a personal vibration plate to take home with them for training which will last for 12 weeks. For the first four weeks, participants will be asked to complete 10 minutes of WBV per day (1 minute on and up to 1 minute of rest), at least 3-4 days per week. At least 24 hours will be recommended in between sessions during weeks 1-4. Beginning at week 5, participants will be asked to increase WBV time to up to 14 minutes and/or reduce the duration of rest. Beginning at week 9, participants will be asked to increase WBV time to up to 20 minutes and/or reduce the duration of rest.

SUMMARY:
The overall goals of this pilot investigation are to determine 1) the feasibility of conducting home based WBV studies, and 2) to determine if sub-acute home based WBV can improve a) exercise capacity, b) conduit- and micro- vascular function, and c) skeletal muscle function.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death in the world and many comorbid conditions (i.e. diabetes, obesity) can affect overall CVD risk. There is increasing interest into the role that skeletal muscle health plays in mediating CVD risk, particularly in metabolic disease states (ie. obesity and diabetes). Whole body vibration (WBV) has emerged as an exercise mimetic that may be more tolerable than traditional modes of exercise, such as treadmill walking/running or cycling. Similar to traditional exercise modalities, WBV can elicit beneficial metabolic effects. In fact, a single bout of WBV increases circulating concentrations of IL-6, which correspond with the normalization of glucose and insulin in obese individuals. The proposed pilot investigation will provide the foundation to begin understanding the molecular and physiological mechanisms of how sub-acute WBV can improve overall CVD risk. We hypothesize that home based WBV will decrease CVD risk by improving skeletal muscle and vascular function via a decrease in systemic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Men and women (> 18 yrs old)
* All races

Exclusion Criteria:

* <18 years old
* Clinical diagnosis of hepatic, cardiovascular, or renal disease
* Diabetic complications (i.e. macrovascular, microvascular, or autonomic)
* Pregnancy
* Direct vasoactive medications (i.e. nitrates)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in VO2 Peak | pre-treatment baseline and following 12 weeks sub-acute whole-body vibration
  change from baseline relative (mL/kg/min) peak oxygen consumption (VO2) during maximal exercise test at 12 weeks
Change in Flow-Mediated Dilation (FMD) | pre-treatment baseline and following 12 weeks sub-acute whole-body vibration
  change from baseline brachial artery flow mediated dilation at 12 weeks.
Change in Skeletal Muscle Mitochondrial Function | pre-treatment baseline and following 12 weeks sub-acute whole-body vibration
  change from baseline skeletal muscle mitochondrial function at 12 weeks. Measured using Near Infrared Spectroscopy (NIRS). Values are an index of phosphocreatine recovery expressed as a rate constant (min-1)
Change in Pulse Wave Velocity (PWV) | pre-treatment baseline and following 12 weeks sub-acute whole-body vibration
  Change from baseline PWV at 12 weeks. Measured by Shygmocor Xcel in m/s.
Change in Post Occlusive Reactive Hyperemia (PORH) | pre-treatment baseline and following 12 weeks sub-acute whole-body vibration
  Change from baseline PORH at 12 weeks. Measured by Laser Speckle Contrast Imager (Moor FLPI).
Change in IL-6 | pre-treatment baseline and following 12 weeks sub-acute whole-body vibration
  change from baseline concentrations of Interleukin 6 (IL-6) obtained via blood draw at 12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University/Georgia Prevention Institute/ Laboratory of Integrative and Exercise Physiology, Augusta, Georgia, United States